CLINICAL TRIAL: NCT05736250
Title: Establishment of a Method for Extraction and Quantification of Gingival Tissue Nicotine in Relation to Conventional Tobacco Biomarkers: a Pilot Study
Brief Title: Establishment of a Method for Extraction and Quantification of Gingival Tissue Nicotine y
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Leila Salhi, PhD, head of clinic, Department of periodontology, buccal surgery and buccal implantology,, University of Liege
Other Study IDs: 2021:250
Record Dates: First submitted 2023-01-24; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Smoking, Cigarette
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TEST group: smoker patients
  Interventions: Diagnostic Test: biopsie

INTERVENTIONS:
Diagnostic Test: biopsie — gingival biopsie

SUMMARY:
establishment of a method for extraction and quantification of gingival tissue nicotine in relation to conventional tobacco biomarkers: a pilot study

DETAILED DESCRIPTION:
The study aim to establish a method for extraction and quantification of gingival tissue nicotine. Additionnaly, the relationship between the nicotine tissue intoxication with others smoking indicators will be evaluated as mentionned in the following PICO question:

* P: Smoker patients
* I: Biopsie of gingival tissue
* C: Non-smoker patient
* O: nicotine dependence test (FTND), salivary cotinine, fibroblast nicotine, number of cigarette consumed per day (NCC) and the pack-year (PY)

ELIGIBILITY:
Inclusion Criteria:

* non smokers
* smokers

Exclusion Criteria:

* not able to have biopsie

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: smoker patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
nicotine | baseline
  nicotine in gingival fibroblast
nicotine dependance | baseline
  Fagerström test for nicotine dependence

SECONDARY OUTCOMES:
salivary cotinine | baseline
number of cigarette consumed | baseline
pack-year | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Salhi, Liège, Liege, Belgium

IPD SHARING:
Plan to Share IPD: No